CLINICAL TRIAL: NCT06747221
Title: HIV Enhanced Access Testing in Emergency Department Program Using a Systems Analysis and Improvement Approach (HEATED-SAIA) Cluster Randomized Trial
Brief Title: Implementation Science to Enhance HIV Testing Services During Emergency Care in Kenya
Acronym: HEATED-SAIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Washington (Other); Brown University (Other)
Responsible Party: Principal Investigator, Adam Aluisio, Associate Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2232153
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: HIV
Keywords: HIV; SAIA; Emergency Care; Africa; Kenya; Emergency Services; HIV Testing Services; Systems Analysis and Improvement Approach; Implementation Science

STUDY DESIGN:
Intervention Model Description: Cluster parallel trial with a baseline measurement period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard care (Active Comparator): Facilities in the control arm will receive regular standard program oversight by county department of health personnel but no further interventions related to the SAIA implementation stratgey.
  Interventions: Other: Systems Analysis and Improvement Approach (SAIA)

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach (SAIA) — SAIA is a 5-step implementation strategy that is repeated every 4-6 weeks for continuous quality improvement. It will be implemented by Kenyan public health workforce and frontline clinical care personnel to systematically identify and address bottlenecks to develop and implement solutions to delivery of HIV Testing Services during emergency department (ED) interactions.
  Step 1: Understanding the cascade of ED patient flow from triage through care conclusion with focus on HTS opportunities. This will support identification of bottlenecks where patients are missed and provides data on potential increases in efficiency if misses are addressed.
  Step 2: Use process mapping to identify modifiable bottlenecks.
  Step 3: Define and implement workflow adaptations to mitigate modifiable bottlenecks.
  Step 4: Monitor changes in performance.
  Step 5: Repeat the analysis and improvement cycle (steps 1-4).

SUMMARY:
There are ~38 million people living with HIV (PLH), with the majority in low-and middle-income countries (LMICs), where the UNAIDS 95-95-95 HIV targets are at risk of not being achieved. Data show that incident infections are concentrated in sub-Saharan Africa and focused in difficult to reach populations. These harder to reach persons frequently also have higher-risk profiles for HIV, making them essential target populations to receive HIV Testing Services (HTS). Among target populations, men, adolescents and young adults (AYAs) aged 15-24 years, and persons from key populations (KPs) represent crucial groups to be reached. In Africa, Emergency Departments (ED) provide care to large numbers of persons that often do not otherwise access health services. Data from Africa show that those seeking emergency care have high burdens of HIV, and desire ED-HTS. As in higher-income countries, EDs in LMICs provide a strategic opportunity to deliver evidence-based HTS interventions to higher-risk persons. In Kenya one in five PLH are unaware of their status, less than half of men are reached for HIV testing at appropriate frequencies, AYAs account for 42% of new infections and KPs contribute to hyper-endemic transmission. To address this, Kenya national strategy calls for utilizing facilities-based care to deliver HTS for difficult to reach populations. However, while the guidelines include EDs as service delivery points, HTS during emergency care in Kenya is still evolving and the evidence-base on best practices is in early development. The HIV Enhanced Access Testing in Emergency Department (HEATED) program in Kenya was developed by a collaborative team led by PI Aluisio (K23AI145411). The HEATED program was derived using the Capability-Opportunity-Motivation Behavioral model to enhance delivery of HTS, through locally appropriate and pragmatic systems initiatives. HEATED program implementation significantly improved HIV testing for the overall ED population by 31%, while also significantly increasing testing for men, AYA and KP and was found to be acceptable by stakeholders. Although pilot evaluation of the HEATED program demonstrated improved HTS for target populations, more robust understanding of optimal implementation strategies in ED settings, impacts on linkage to HIV care outcomes, costing and maintenance data are needed to inform development of ED-HTS programming in Kenya. To address this, the current proposal will build upon the HEATED program by evaluating use of the Systems Analysis and Improvement Approach (SAIA) implementation strategy (HEATED-SAIA) to improve HTS in a cluster randomized trial in all Ministry of Health EDs in Kilifi, Mombasa and Kwale Counties of the Coast Region of Kenya. The Reach, Effectiveness, Adoption, Implementation and Maintenance framework with quantitative and qualitative data will be used in trial assessment. Building on the K23 pilot data and leveraging SAIA, the HEATED-SAIA program has substantial potential to improve HTS delivery by strategically and pragmatically engaging difficult to reach populations already interfacing with emergency health systems, while being acceptable and cost-effective.

DETAILED DESCRIPTION:
Globally, there are ~38 million people living with HIV (PLH), with the majority in low-and middle-income countries (LMICs), where the UNAIDS 95-95-95 HIV targets are at risk of not being achieved. Data show that incident infections are concentrated in sub-Saharan Africa (SSA) and focused in difficult to reach populations for HIV services. These persons also often have higher-risk profiles for HIV making them priority populations to receive HIV Testing Services (HTS). Among target populations, men, adolescents and young adults (AYAs) aged 15-24 years, and persons from key populations (KPs), are crucial groups which must be regularly reached for HTS to achieve global control targets.

In LMICs, emergency departments (ED) provide care to large numbers of persons that often do not otherwise access health services. Injuries among men, AYA and KPs are frequent reasons for ED care. Data from Africa show that persons seeking emergency care have high HIV burdens, and desire ED-HTS. Furthermore, as EDs are status-neutral care settings, ED-HTS may have fewer stigmatization barriers than conventional service delivery points (SDPs) to support testing provision. However, data from multiple SSA studies show that ED HIV testing is infrequent, with <25% of patients engaged for HTS during emergency care. EDs in LMICs represent a waiting strategic and pragmatic opportunity to deliver evidence-based HTS to higher-risk persons already frequently in contact with health facilities.

While Kenya has reduced its HIV prevalence to ~4.0%, incidence reduction targets have not been met, and in 2021 there was an 7.8% increase in new infections. In Kenya, one in five people with HIV disease are undiagnosed, less than half of men are reached for HIV testing at appropriate frequencies, AYAs account for 42% of new infections and KPs contribute to hyper-endemic transmission. Kenya's national guidelines call for utilizing facilities-based care to deliver HTS for difficult to reach populations where the HIV epidemic is concentrated. While the guidelines include EDs as SDPs, emergency care HTS is still evolving in Kenya and best practice evidence is in early development. The HIV Enhanced Access Testing in Emergency Departments (HEATED) program in Nairobi, Kenya was developed by a collaborative team led by Principal Investigator (PI) Dr. Aluisio (K23AI145411). The program was a status neutral systems intervention, using the Capability-Opportunity-Motivation Behavioral model to enhance ED-HTS, through data-driven, setting-specific, feasible systems adaptations designed to address modifiable barriers (micro-strategies). The HEATED program significantly improved likelihood of ED-HTS for the overall population by 31%, and significantly increased testing for men, AYA and KP. In addition, stakeholders affirmed that the program was acceptable.

Although evaluation of the HEATED program demonstrated improved HTS more robust understanding of optimal implementation strategies, impacts on linkage to HIV care and costing data are needed to inform ED-HTS advancement in Kenya. To address this, the current proposal builds upon the HEATED program by utilizing and evaluating the Systems Analysis and Improvement Approach (SAIA) implementation strategy (HEATED-SAIA) to enhance HTS delivery in a cluster randomized trial of all public facilities with EDs in Kilifi, Mombasa and Kwale Counties of the Coast region of Kenya. SAIA is a multi-component implementation strategy that utilizes cascade analysis, process flow mapping and micro-strategy development and testing in plan-do-study-act cycles to improve care delivery.46 SAIA implementation has been shown to improve HTS integration in family planning (FP) clinics in Mombasa County by the study team previously. Application of SAIA to ED settings in the Coast region has substantial potential to improve delivery of evidence-based HTS for higher-risk persons already in contact with care, while also expanding the evidence-base for SAIA via application in a novel clinical space. This will be studied through the following aims:

Aim 1: Evaluate impacts of the HEATED-SAIA program as compared to standard care (control) in a cluster randomized trial of all ten public ED facilities in three counties in the Coast region of Kenya, to improve HIV screening, testing, and linkage to treatment and prevention, among persons receiving emergency care with a focus on target populations of men, AYA and KPs.

Approach: This cluster parallel trial, with a baseline measurement period, will randomize all ten public EDs in Kilifi, Mombasa and Kwale Counties (1:1) to control (usual care) or intervention (SAIA implementation strategy) and use the Reach, Effectiveness, Adoption, Implementation and Maintenance (REAIM) framework in trial assessment. Quantitative systems level data and qualitative participant level data, based on the Consolidated Framework for Implementation Research and the Implementation Research Logic Model will be used to inform appropriate use of the results in the study setting and larger public health context of Kenya.

Aim 2: Assess the cost of ED-HTS and implementation of the HEATED-SAIA program using micro-costing and time-and-motion costing methods to inform public health programming and future scale-up.

ELIGIBILITY:
Facility Level (Quantitative De-identified Systems Data)

Inclusion Criteria:

* Kenya public health facilities in Kwale, Mombassa and Kilifi Counties
* Have an active emergency department
* Have HIV testing services either embedded in the emergency department or the facility.

Exclusion Criteria:

* Private health facilities
* Kenya public health facilities in Kwale, Mombassa and Kilifi Counties without an active emergency department
* Kenya public health facilities in Kwale, Mombassa and Kilifi Counties without existing HIV testing services

Participant Level (Qualitative Data) Healthcare Personnel

Inclusion Criteria:

* Personnel working at the departments of health in Kwale, Mombassa and Kilifi Counties
* Personnel working at a Kenya public health facilities randomized to the control or intervention arm in Kwale, Mombassa and Kilifi Counties
* Age 18 years or greater
* Able and willing to provide informed consent

Exclusion Criteria:

* Personnel not working at a Kenya public health facilities randomized to the control or intervention arm in Kwale, Mombassa and Kilifi Counties
* Age less than 18 years
* Not able and willing to provide informed consent

Participant Level (Qualitative Data) ED-HTS Clients

Inclusion Criteria:

* Patients receiving emergency care and engaged for ED-HTS at a Kenya public health facilities randomized to the intervention arm of the trial in Kwale, Mombassa and Kilifi Counties
* Age 18 years or greater
* Able and willing to provide informed consent

Exclusion Criteria:

* Age less than 18 years
* Not able and willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Reach: Staff Engagement | Quarterly (3-42 months)
  1. Proportion of personnel taking part in SAIA cycles (intervention sites)
  2. Representativeness of staff taking part in SAIA cycles planning (intervention sites)
Reach: Patient Participation | Quarterly (3-42 months)
  1. Proportion of ED patients accepting referral for HTS among those screened & eligible (intervention versus control sites)
  2. Proportion of ED patients accepting referral for HTS for target populations of men and AYA among those screened & eligible (intervention versus control sites)
Effectiveness: HIV Testing Delivery | Quarterly (3-42 months)
  1. Proportion of ED patients completing testing among patients appropriate for testing (intervention versus control sites)
  2. Proportion of ED patients completing testing among target populations men and AYA appropriate for testing (intervention versus control sites)
  3. Proportion of ED persons from KPs completing testing (intervention versus control sites)
Effectiveness: Linkage to Care for People Living with HIV | Quarterly (3-42 months)
  1. Proportion of ED patients tested identified as PLH linked to HIV care (intervention versus control sites)
  2. Proportion of ED patients tested identified as PLH linked to HIV care among target populations of men and AYA (intervention versus control sites)
  3. Proportion of ED persons from KPs tested identified as PLH linked to HIV care (intervention versus control sites)
Effectiveness: PrEP Screening & Referral | Quarterly (3-42 months)
  1. Proportion of ED patients testing negative screened and referred for PrEP (intervention versus control sites)
  2. Proportion of ED patients testing negative among target populations of men and AYA screened and referred for PrEP (intervention versus control sites)
  3. Proportion of ED persons from KPs testing negative screened and referred for PrEP (intervention site versus controls)
Adoption: Uptake Determinants | Months: 1, 3 & 15
  IRLM-CFIR qualitative data to understand HEATED-SAIA determinants of uptake (Primary SAIA Facilitators, Primary SAIA Implementers, DOH Personnel)
Adoption: Staff Intentions | Months: 1, 6, 9 & 15
  CPD-reaction assessments for ED and HTS personnel on HEATED-SAIA program (intervention sites)
Implementation: Feasibility | Monthly (3-42 months)
  1. Proportion of micro-strategies/cycle delivered subsequent cycle (intervention sites)
  2. Proportion of micro-strategies identified and adopted from all HEATED-SAIA cycles delivered in the facility for >6 months (intervention sites)
  3. Integrated IRLM-CFIR qualitative data & coincidence analysis of micro-strategies (intervention sites)
Implementation: Fidelity | Months: 3, 15, & 40
  Qualitative data using IRLM-CFIR to understand HEATED-SAIA cycle fidelity (Primary SAIA Implementers at intervention site) (intervention sites)
Implementation: Facilitators & Barriers | Months: 3, 15, 24 & 40
  IRLM-CFIR qualitative data on facilitators and barriers of HEATED-SAIA cycle completion (Primary SAIA Facilitators, Primary SAIA Implementers, DOH Personnel, ED-HTS clients)
Maintenance: Sustainability | Months: 24, 30, 36 & 42
  1. Continuation of HEATED-SAIA cycles with >3 per 6 months (intervention site)
  2. IRLM-CFIR qualitative data to understand determinates of HEATED-SAIA continuation in the absences of research staff (Primary SAIA Facilitators, Primary SAIA Implementers, DOH Personnel, ED-HTS clients)
Maintenance: Penetration | Months: 24 & 40
  Quantitative and qualitative data (IRLM-CFIR) to understand integration of HEATED-SAIA into institutional policy and procedures and related determinates for integration (Primary SAIA Facilitators, Primary SAIA Implementers, DOH Personnel)
Economic evaluation: ED-HTS and implementation of the HEATED-SAIA program | months 3, 15 & 21
  Micro-costing and time-and-motion costing for ED-HTS programing (baseline) and HEATED-SAIA programming

IPD SHARING:
Plan to Share IPD: Undecided